CLINICAL TRIAL: NCT06995248
Title: Effect of Laughter Yoga on Pain, Fatigue and General Well-Being in Cancer Patients and Their Caregivers: A Randomized Controlled Study
Brief Title: The Effect of Laughter Yoga on Pain, Fatigue, and General Well-Being in Cancer Patients and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Birim Kiper, nurse, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0009000956254142
Record Dates: First submitted 2025-05-10; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Laughter Yoga
Keywords: pain; caregives; fatigue; laughter therapy; cancer patients
MeSH Terms: conditions — Pain; Fatigue | interventions — Laughter Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter Yoga Group (Experimental): Participants in this group will receive a 6-session laughter yoga program over a 2-week period. Each session includes breathing exercises, intentional laughter practices, and light physical activity. The intervention is designed to reduce stress, enhance well-being, and improve pain and fatigue levels.
  Interventions: Behavioral: Laughter Yoga
- control arm (No Intervention): Participants in this group will not receive any behavioral intervention during the study period. They will only complete the pre- and post-assessment questionnaires at the same intervals as the experimental group, allowing for outcome comparison.

INTERVENTIONS:
Behavioral: Laughter Yoga — Laughter yoga sessions are a behavioral intervention regularly conducted to help participants reduce stress, build social connections, and enhance overall well-being.
  Arms: Laughter Yoga Group

SUMMARY:
This study aims to evaluate the effect of laughter yoga on pain, fatigue, and general well-being in cancer patients and their caregivers. Participants will be randomly assigned to either a laughter yoga intervention group or a control group. The intervention group will receive six sessions of laughter yoga over two weeks. Outcomes will be measured before and after the intervention.

DETAILED DESCRIPTION:
Laughter yoga is a complementary mind-body practice that combines unconditional laughter with breathing techniques. It has been shown to reduce stress, improve mood, and promote psychological and physiological well-being. This randomized controlled trial will assess the effectiveness of a 6-session laughter yoga program on reducing pain and fatigue and enhancing general well-being in cancer patients and their caregivers. Participants in the experimental group will attend three sessions per week for two weeks, each lasting approximately 30-40 minutes. Outcomes will be measured before and after the intervention using validated scales.

Pain will be assessed using the Visual Analog Scale (VAS), which measures pain intensity on a scale from 0 (no pain) to 10 (worst possible pain).

Fatigue will be measured using the Visual Analogue Scale for Fatigue (VAS-F), a validated instrument that evaluates the intensity of fatigue and its impact on daily activities.

The General Well-Being Scale is a self-report instrument used to assess an individual's overall psychological well-being.he scale includes items related to mood, emotional state, and general life satisfaction. It is typically measured using a Likert-type format, where participants rate the frequency and intensity of their feelings or experiences on a scale (e.g., from "strongly disagree" to "strongly agree").

These validated scales will be administered at baseline (before the intervention) and at the end of the intervention (after the 6 sessions) to assess changes in the primary outcomes of pain, fatigue, and general well-being.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who volunteer to participate in the study

Exclusion Criteria:

* having asthma or COPD
* being under 18 or over 65 years of age, and having any health condition or disability that impairs communication (such as visual or hearing impairments, or neurological or psychiatric disorders).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-09-02 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Level | Before and one week after the 6-session laughter yoga program
  Pain will be measured using the Visual Analog Scale (VAS) at baseline and one week after the final session to assess the effectiveness of the intervention.

SECONDARY OUTCOMES:
Change in Fatigue Level | Before the intervention and one week after
  Change in fatigue level measured by the Visual Similarity Scale for Fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morishima T, Miyashiro I, Inoue N, Kitasaka M, Akazawa T, Higeno A, Idota A, Sato A, Ohira T, Sakon M, Matsuura N. Effects of laughter therapy on quality of life in patients with cancer: An open-label, randomized controlled trial. PLoS One. 2019 Jun 27;14(6):e0219065. doi: 10.1371/journal.pone.0219065. eCollection 2019. PMID 31247017